CLINICAL TRIAL: NCT03578939
Title: Next Generation Sequencing di Cellule Tumorali Nell'Adenocarcinoma Pancreatico Localmente Avanzato
Brief Title: Next Generation Sequencing of Tumor Cells in Locally Advanced Pancreatic Adenocarcinoma
Acronym: LAPC-NGS-A/001
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 1890
Record Dates: First submitted 2018-02-19; First posted 2018-07-06 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Biopsy EUS guided — NGS Sequencing on Biopsy samples

SUMMARY:
All patients referring to the U.O .of Digestive Endoscopy of the Humanitas Hospital to undergo EUS with biopsy in the pre-treatment evaluation of locally advanced pancreatic adenocarcinoma, satisfying all the inclusion criteria and without any of the exclusion criteria, will be enrolled.

Patients will then undergo endoscopic procedures (EUS with biopsy) provided by good clinical practice in consideration of the suspected diagnosis for which they come to Investigator's attention.

Biopsy will be performed using a histology needle (22 G, Acquire, Boston Scientific, MA, United States). The obtained material will be processed in the Pathological Anatomy. A small part of this will be sent to the NGS analysis.

At the time of preparation for the examination, the patients will be asked for blood collection (10 ml of blood) in order to evaluate any circulating tumor cells that will be identified by SmartBioSurface technique (Tethis S.p.A) and analyzed by appropriate molecular markers and NGS.

The clinical evaluation of the patient will take place at 6 months from the date of the procedure, through telephone contact and / or outpatient visit.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years,
* Signature of informed consent,
* Naïve patients with pancreatic adenocarcinoma (confirmed cito/ histologically), not subjected to previous treatments,
* Need to perform EUS with biopsy,
* Life expectancy over 6 months.

Exclusion Criteria:

* Patients with non-primary pancreatic tumors, pancreatic neuroendocrine tumors or benign pancreatic masses
* Patients who have already undergone cancer treatment of any kind

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients belonging to the U.O. of Digestive Endoscopy of the Humanitas Hospital to undergo EUS with biopsy in the pre-treatment evaluation of locally advanced pancreatic adenocarcinoma.
  At the time of preparation for the examination, patients will be asked for blood collection (10 ml of blood) in order to evaluate any circulating tumor cells.
  Patients will then be subjected to the endoscopic procedure (EUS with biopsy) provided for by good clinical practice in consideration of the suspected diagnosis for which they come to our attention.
Sampling Method: Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Isomatic genetic mutations will be evaluated in locally advanced naïve pancreatic adenocarcinoma in order to better understand the best way to treat patient. | 18 Months

SECONDARY OUTCOMES:
Adequacy of samples obtained by biopsy - EUS guided with needles Acquire from 22G in providing the diagnosis, | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Carrara, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrara S, Solda G, Di Leo M, Rahal D, Peano C, Giunta M, Lamonaca L, Auriemma F, Anderloni A, Fugazza A, Maselli R, Malesci A, Laghi L, Repici A. Side-by-side comparison of next-generation sequencing, cytology, and histology in diagnosing locally advanced pancreatic adenocarcinoma. Gastrointest Endosc. 2021 Mar;93(3):597-604.e5. doi: 10.1016/j.gie.2020.06.069. Epub 2020 Jul 5. PMID 32640200